CLINICAL TRIAL: NCT04555122
Title: COVID-19 Ad Intervention for Social Distancing
Brief Title: COVID-19 Ad Intervention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Per Sponsor Request; nonACT
Sponsor: University of California, Irvine (Other)
Collaborators: City University of Hong Kong (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Sean D Young, Associate Professor of Emergency Medicine and Informatics, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB# 20205923
Record Dates: First submitted 2020-04-29; First posted 2020-09-18 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Social Distance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Advertisements will be sent to participants to attempt to increase adherence to stay-at-home orders and social distancing. There are 3 types of advertisements. This will occur for 7 days.
  Interventions: Behavioral: Social Distancing Advertisements
- Control Group (No Intervention): Control Group will be people who will not receive any advertisements.

INTERVENTIONS:
Behavioral: Social Distancing Advertisements — Participants will receive 3 types of advertisements to increase social distancing/staying at home.
  Arms: Intervention Group

SUMMARY:
This study will provide advertisements to (de-identified) participants and track (de-identified) movement patterns to learn whether the ads increase adherence to stay-at-home orders.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older (as identified by company running advertisements); recent visit to a non-essential location; agreed to terms and conditions of websites allowing advertisements

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-05-28 (Estimated); Study Completion 2022-07-28 (Estimated)

PRIMARY OUTCOMES:
Mobility | 7 days
  Amount of time that participants are outside of their primary location/home

CONTACTS AND LOCATIONS:
Locations (1):
- UC Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No